CLINICAL TRIAL: NCT00005042
Title: A Multicenter, Open-Label, Phase II Study of SU5416 in Patients With Cutaneous AIDS-Related Kaposi's Sarcoma
Brief Title: SU5416 in Treating Patients With AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: AMC-022; CDR0000067633 (Other: NCI); NCT00005932 (obsolete NCT alias)
Record Dates: First submitted 2000-04-06; First posted 2004-07-19 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Sarcoma
Keywords: AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi | interventions — Semaxinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: semaxanib

SUMMARY:
RATIONALE: SU5416 may stop the growth of Kaposi's sarcoma by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of SU5416 in treating patients who have AIDS-related Kaposi's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antitumor effects of SU5416 in patients with chemotherapy refractory cutaneous AIDS-related Kaposi's sarcoma. II. Determine the safety and tolerability of this regimen in these patients. III. Determine the pharmacokinetics of this regimen in these patients. IV. Determine the safety of this regimen on HIV replication and immune parameters in these patients. V. Determine the effects of this regimen on overall quality of life and tumor specific symptoms in these patients.

OUTLINE: This is a multicenter study. Patients receive SU5416 IV twice weekly for 4 weeks. Treatment continues for up to 1 year in the absence of disease progression or unacceptable toxicity. Quality of life is assessed. Patients are followed at 30 days after the last treatment, and every 3 months thereafter.

PROJECTED ACCRUAL: A total of 29 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, cutaneous AIDS-related Kaposi's sarcoma (KS) Must have failed at least 1 standard chemotherapy regimen for KS Chemotherapy refractory (progressed during anthracycline-based or paclitaxel therapy) OR Chemotherapy intolerant (hypersensitivity to drug or unacceptable toxicity) HIV positive At least 5 measurable cutaneous lesions No prior radiotherapy or intradermal therapy to indicator lesions OR KS-related generalized edema or edema of the extremities without evidence of active cutaneous lesions

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 50-100% Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 500/mm3 Platelet count at least 50,000/mm3 Hepatic: AST no greater than 5.0 times upper limit of normal Bilirubin no greater than 2.0 mg/dL (no greater than 3.0 mg/dL if concurrent indinavir therapy) Renal: No history of renal failure Creatinine no greater than 1.8 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No myocardial infarction within the past year No severe or unstable angina No history of unstable atherosclerotic coronary artery disease requiring coronary or peripheral artery bypass surgery within the past 2 years Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No known hypersensitivity to Cremophor or Cremophor based drug product No uncontrolled serious infection such as: Pneumocystis carinii pneumonia Toxoplasmic brain abscess CMV retinitis or colitis Cryptococcal meningitis Symptomatic Mycobacterium avium-intracellulare No other active malignancy, except: Basal cell skin cancer Carcinoma in situ of the cervix No cerebral bleed No diabetes mellitus with clinical evidence of severe peripheral vascular disease or diabetic ulcers No other acute or chronic medical or psychiatric condition that would preclude compliance No history of metabolic acidosis from nucleoside analogues Anion gap no greater than 11 (Na - Cl, HCO3)

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 2 weeks since prior immunotherapy for AIDS-related KS and recovered At least 2 weeks since prior biologic therapy for AIDS-related KS No concurrent immunotherapy Chemotherapy: See Disease Characteristics At least 2 weeks since prior chemotherapy for AIDS-related KS and recovered No other concurrent systemic chemotherapy Endocrine therapy: At least 2 weeks since prior hormonal therapy for AIDS-related KS No concurrent hormonal therapy (including beta-HCG) Radiotherapy: See Disease Characteristics At least 2 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: At least 4 weeks since prior surgery No prior stereotactic surgery Other: Stable antiretroviral therapy for at least 4 weeks prior to and at least 29 days during the study Concurrent FDA approved antiretroviral agents or expanded access antiretroviral agents allowed At least 3 weeks since other prior investigational agents No concurrent local or topical therapy for AIDS-related KS No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Miles, MD, Study Chair — UCLA Clinical AIDS Research and Education (CARE) Center
Locations (2):
- United States (2):
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York